CLINICAL TRIAL: NCT05016700
Title: Correlation of Clinical Symptoms With Neuromorphological Changes of the Colorectal Wall in Patients With a Bowel Evacuation Disorder
Brief Title: Neuropathological Changes of the Intestinal Wall in Patients With Bowel Evacuation Disorders
Acronym: Constipation
Status: Recruiting | Type: Observational
Sponsor: Evangelisches Klinikum Köln Weyertal gGmbH (Other)
Collaborators: University of Cologne (Other)
Responsible Party: Principal Investigator, Claudia Rudroff, Head of the Department of Visceral Surgery and Functional Surgery of the lower GI Tract, Evangelisches Klinikum Köln Weyertal gGmbH
Other Study IDs: EVKKoeln
Record Dates: First submitted 2021-07-24; First posted 2021-08-23 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Defecation Disorder; Neuropathology; Autoimmune Diseases
Keywords: Neuropathology; Defecation disorder; Autoimmune disease; Hypoganglionosis; Autoimmune ganglionitis; Neurological bowel disorder; Colon surgery
MeSH Terms: conditions — Autoimmune Diseases | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Blood samples (EDTA) to investigate immunological activation for the individual patient
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: blood sample — we want to identify a diagnostic option to identify patients, who have a neuropathological distraction of their ganglia cells in the bowel

SUMMARY:
Constipation and defecation disorders affect about 15% of the European population and of those up to 30% of the patients over 65 years of age. For those affected, this is associated with major restrictions in quality of life and high health care costs .

The underlying causes of constipation and defecation are complex and only partially understood.

Intestinal (full wall) resections taken in clinical practice from these patients when conservative therapy has been exhausted show rarefaction of ganglion cell nests in the myenteric plexus and submucosal plexus as well as changes in cholinergic innervation.

Initial histopathological investigations suggest an inflammatory genesis of this rarefaction of ganglion cell nests, which will be further characterised/investigated in the context of this study on the basis of further histopathological and serological investigations. This may lead to novel therapeutic approaches that can causally treat the symptoms of those affected.

DETAILED DESCRIPTION:
Intestinal transit disorders (constipation/obstipation) and/or defecation disorders (expulsion disorders) are widespread symptoms in our culture, which, depending on their severity, can become a disease. Epidemiological studies show that up to 30% of the population over the age of 65 is affected. The suffering of those affected is usually very high.

The patients are usually treated conservatively at first. The focus is on lifestyle changes, dietary adjustments and medication to support bowel movements. If the symptoms persist despite consistent conservative therapy, additional diagnostics such as laboratory tests, sonography and colonoscopy are performed.

Further diagnostic steps include anal manometry, defecography and colon transit time.

From 2015 onwards, the systematic neuropathological examination of whole-wall samples was performed on the bowel specimen of patients who were surgically treated for defecation disorders. In addition, in individual cases in which no bowel resection was indicated, rectal full-wall samples were taken to confirm the diagnosis and indication for sacral nerve stimulation (SNS) and examined neuropathologically in the same way. The intestinal wall was examined for ganglion cell nests in the myenteric plexus and the submucosal plexus in order to identify the pathophysiological cause of the transport disorder.

The analysis showed rarefaction of the ganglion cell nests in the myenteric plexus and the submucosal plexus, as well as both a change in the cholinergic innervation and changes that suggest an autoimmune initiated process.

Increasing evidence links gastroenteritic germs with chronic intestinal motility disorders, so that a Campylobacter or Yersinia infection could well be the trigger for the observed neuropathological changes.

The aim of the study is to analyse the pathomechanism of chronic intestinal emptying disorders. Neuropathological findings on the plexus of the intestinal wall specimen are correlated to clinical findings measured by clinical scores in order to identify a diagnostic pattern.

ELIGIBILITY:
Inclusion Criteria:

* obstructive defecation disorder scheduled for surgery
* must be able to undergo surgery
* > 18 years of age
* informed consent

Exclusion Criteria:

* no defecation disorder
* no surgery needed
* unable to undergo surgery
* ≤ 18 years
* no consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with severe defecation disorders, both in terms of colonic transit disorder and obstructive defecation disorder, and combinations of both, who have been managed conservatively and require a full-wall bowel biopsy or bowel resection for medical indication.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2019-03-20 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2033-12-31 (Estimated)

PRIMARY OUTCOMES:
Neuropathological changes of the intestinal wall in patients with bowel evacuation disorder in correlation to clinical defecation score | 10 years
  Clinical outcome measure by score: Altomare Score (name of initiator) score (minimum 0 to maximum 30 points; higher values mean worse outcome)

SECONDARY OUTCOMES:
Correlation of psychic health and neuropathological changes of the intestinal wall in patients with defecation disorder | 10 years
  Changes in QoL and relief from depressive symptoms after surgery measured by clinical psysic health questionnaire (PHQ 9) ; minimum 0 to maximum 27 points; higher scores mean worse outcome
Correlation of anxiety scoring and neuropathological changes of the intestinal wall in patients with defecation disorder | 10 years
  Changes in anxiety symptoms after surgery measured by clinical general anxiety score (GAD 7); minimum 0 to maximum 21 points; higher scores mean worse outcome
Association of pathological findings for autoimmune activation with duration of symptoms according to medical history | questionaire at inclusion to study
  Onset of symptoms in correlation to severity and picture of pathological findings in months
Association of pathological findings for autoimmune reaction with an initiating event according to the medical questionaire | questionaire at inclusion to study
  Identification of an initiating event to the occurrence of the symptoms
Correlation of abdominal discomforting symptoms and neuropathological changes of the intestinal wall in patients with bowel evacuation disorder | 10 years
  Clinical outcome measure rectal toxicity score (minimum 0 to maximum 32 points; higher scores mean worse outcome)
Correlation of neuropathological changes of the intestinal wall in patients with bowel evacuation disorder and clinical defecation insufficiency (incontinence) | 10 years
  Clinical outcome measure by score: Wexner (name of initiator) incontinence score (minimum 0 to maximum 20 points; higher scores mean worse outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Rudroff, MD, Principal Investigator — Claudia Rudroff, MD PhD
Locations (1):
- Evangelisches Klinikum Koeln Weyertal, Cologne, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: Yes
After publication of data all data will be uploaded to clinical trials
Supporting Information: Study Protocol, ICF
Time Frame: now
Access Criteria: open

REFERENCES:
- [Background] Han EC, Oh HK, Ha HK, Choe EK, Moon SH, Ryoo SB, Park KJ. Favorable surgical treatment outcomes for chronic constipation with features of colonic pseudo-obstruction. World J Gastroenterol. 2012 Aug 28;18(32):4441-6. doi: 10.3748/wjg.v18.i32.4441. PMID 22969211
- [Background] Bassotti G, Villanacci V, Nascimbeni R, Asteria CR, Fisogni S, Nesi G, Legrenzi L, Mariano M, Tonelli F, Morelli A, Salerni B. Colonic neuropathological aspects in patients with intractable constipation due to obstructed defecation. Mod Pathol. 2007 Mar;20(3):367-74. doi: 10.1038/modpathol.3800748. Epub 2007 Feb 2. PMID 17277762
- [Background] Bassotti G, Villanacci V, Cathomas G, Maurer CA, Fisogni S, Cadei M, Baron L, Morelli A, Valloncini E, Salerni B. Enteric neuropathology of the terminal ileum in patients with intractable slow-transit constipation. Hum Pathol. 2006 Oct;37(10):1252-8. doi: 10.1016/j.humpath.2006.04.027. Epub 2006 Jul 20. PMID 16949932
- [Background] Bassotti G, Villanacci V, Maurer CA, Fisogni S, Di Fabio F, Cadei M, Morelli A, Panagiotis T, Cathomas G, Salerni B. The role of glial cells and apoptosis of enteric neurones in the neuropathology of intractable slow transit constipation. Gut. 2006 Jan;55(1):41-6. doi: 10.1136/gut.2005.073197. Epub 2005 Jul 24. PMID 16041063
- [Background] Wedel T, Roblick UJ, Ott V, Eggers R, Schiedeck TH, Krammer HJ, Bruch HP. Oligoneuronal hypoganglionosis in patients with idiopathic slow-transit constipation. Dis Colon Rectum. 2002 Jan;45(1):54-62. doi: 10.1007/s10350-004-6114-3. PMID 11786765
- [Background] Valli PV, Pohl D, Fried M, Caduff R, Bauerfeind P. Diagnostic use of endoscopic full-thickness wall resection (eFTR)-a novel minimally invasive technique for colonic tissue sampling in patients with severe gastrointestinal motility disorders. Neurogastroenterol Motil. 2018 Jan;30(1). doi: 10.1111/nmo.13153. Epub 2017 Jul 6. PMID 28681569
- [Background] Do MY, Myung SJ, Park HJ, Chung JW, Kim IW, Lee SM, Yu CS, Lee HK, Lee JK, Park YS, Jang SJ, Kim HJ, Ye BD, Byeon JS, Yang SK, Kim JH. Novel classification and pathogenetic analysis of hypoganglionosis and adult-onset Hirschsprung's disease. Dig Dis Sci. 2011 Jun;56(6):1818-27. doi: 10.1007/s10620-010-1522-9. Epub 2011 Jan 11. PMID 21222160
- [Background] Porter CK, Choi D, Cash B, Pimentel M, Murray J, May L, Riddle MS. Pathogen-specific risk of chronic gastrointestinal disorders following bacterial causes of foodborne illness. BMC Gastroenterol. 2013 Mar 8;13:46. doi: 10.1186/1471-230X-13-46. PMID 23510245
- [Background] Mearin F, Perello A, Balboa A, Perona M, Sans M, Salas A, Angulo S, Lloreta J, Benasayag R, Garcia-Gonzalez MA, Perez-Oliveras M, Coderch J. Pathogenic mechanisms of postinfectious functional gastrointestinal disorders: results 3 years after gastroenteritis. Scand J Gastroenterol. 2009;44(10):1173-85. doi: 10.1080/00365520903171276. PMID 19711225
- [Result] Sanchez-Ruiz M, Brunn A, Montesinos-Rongen M, Rudroff C, Hartmann M, Schluter D, Pfitzer G, Deckert M. Enteric Murine Ganglionitis Induced by Autoimmune CD8 T Cells Mimics Human Gastrointestinal Dysmotility. Am J Pathol. 2019 Mar;189(3):540-551. doi: 10.1016/j.ajpath.2018.11.016. Epub 2018 Dec 27. PMID 30593823

DOCUMENTS (2):
  • Study Protocol (2018-10-18): https://cdn.clinicaltrials.gov/large-docs/00/NCT05016700/Prot_000.pdf
  • Informed Consent Form (2019-02-27): https://cdn.clinicaltrials.gov/large-docs/00/NCT05016700/ICF_001.pdf